CLINICAL TRIAL: NCT03244891
Title: Effects of Low Central Volume and Intermittent Positive Pressure Ventilation on the Heart Rate Variability
Brief Title: Autonomic Challenges From Mild Hypovolemia and Mechanical Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ASST Fatebenefratelli Sacco (Other)
Responsible Party: Principal Investigator, Riccardo Colombo, Principal Investigator, ASST Fatebenefratelli Sacco
Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: HRV2017_Healthy
Record Dates: First submitted 2017-08-05; First posted 2017-08-10 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Autonomic Nervous System Imbalance; Hypovolemia; Positive-Pressure Respiration
MeSH Terms: conditions — Hypovolemia | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Studied subjects (Experimental): Each subject will be studied during two sequential phases:
  1. before fluid challenge
  2. after fluid challenge
  During each phase, the subjects will be studied at:
  1. baseline - spontaneously breathing
  2. head down position - spontaneously breathing
  3. baseline - positive pressure ventilation
  4. head down position - positive pressure ventilation The sequence a-b-c-d will be randomized for each subject and for each phase
  Interventions: Other: Increase of central volume; Other: Ventilation mode

INTERVENTIONS:
Other: Increase of central volume — Mild hypovolemia will be induced in healthy volunteers by 12 hours fasting. Three conditions will be considered for the analysis, each of them both during spontaneous breathing and positive pressure ventilation:
  1. baseline
  2. after fluid shift induced by passive head down position at 15 degrees
  3. after fluid challenge with Ringer acetate 15ml*kg in head down position
  A total of six steps will be considered for the analysis
Other: Ventilation mode — Each previous step will be done in two respiratory conditions:
  1. spontaneous breathing
  2. noninvasive ventilation via facial mask in pressure support mode at 8 cmH2O above positive end expiratory pressure of 5 cmH2O, inspiratory fraction of oxygen of 0.25 In both conditions respiratory rate will be set at 18 breaths per min following a metronome

SUMMARY:
Heart Rate Variability (HRV) analysis has been studied in the critically ill patients although it is affected by several uncontrolled variables in the clinical conditions. The aim of this trial is to measure the effects of mildly reduced central volume and cyclic variation of intrathoracic pressure on the variables frequently used to describe the HRV.

DETAILED DESCRIPTION:
Twelve healthy volunteers will be studied. Mild hypovolemia will be induced by 12 hours fasting from food and drinks. At 8.30 AM the study protocol will start. The studied subjects will lie calm supine in a ICU bed able to provide passive head up and head down tilt. They will be connected to a Siemens SC9000 monitor showing their ECG waves and to a Nexfin (BMEYE) monitor for continuous noninvasive blood pressure (NBP) assessment. Both waves (ECG and NBP) will be recorded on a laptop PC through analogic/digital input/output converter (PowerLab 8/35, ADinstruments). The studied subjects will undergo to a sequence of (1) spontaneous breathing at 10 degrees head up, (2) spontaneous breathing at 7 degrees head down, (3) noninvasive ventilation at 10 degrees head up, and (4) noninvasive ventilation at 7 degrees head down. The sequence 1-2-3-4 will be randomized. After this four phases, a fluid challenge of ringer acetate 15ml*kg will be intravenously administered and the a sequence 1-2-3-4 will be repeated after a new randomization. Noninvasive ventilation will be provided with a facial mask with ventilatory setting: Psupp 8 cmH2O, PEEP 5 cmH2O, FiO2 0.28. Psupp will be decreased by 2 cmH2O steps if the inspiratory tidal volume will be >10ml*kg. During both spontaneous breathing and noninvasive ventilation the subjects will breathe following a metronome at 18bpm.

HRV analysis will be conducted following the recommendation of the Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology (see reference).

Furthermore, the healthy volunteers will be studied by trans-thoracic ultrasound assessment with a Philips EPIQ7 sonographer, during each study phase.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* history of cardiac, metabolic, respiratory, renal, neurological or hematologic disease of any kind
* chronically assuming drugs of any kind
* non sinus cardiac rhythm
* ectopic beats >5% of all cardiac beats
* claustrophobia or unable to tolerate noninvasive ventilation via facial mask

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Effects of increasing central blood volume on heart rate variability | 10 mins each step
  The studied subjects will undergo to increase of central blood volume in two steps:
  1. passive head down tilt at -7 degrees
  2. intravenous infusion of ringer acetate of 15ml*kg body weight
Effect of cyclic intrathoracic pressure oscillations on heart rate variability | 10 min each step
  The studied subject will undergo to two ventilatory modes:
  1. spontaneous breathing at 18 breaths per min
  2. positive pressure ventilation via face mask

SECONDARY OUTCOMES:
Effects of increasing central blood volume and of cyclic intrathoracic pressure oscillations on echographic cardiac function variables | 10 mins each step
  At each step cardiac functionality assessment will be done by transthoracic echocardiography

CONTACTS AND LOCATIONS:
Locations (1):
- ASST Fatebenefratelli Sacco, Luigi Sacco Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guyton JE, Arthur C. The Autonomic Nervous System and The Adrenal Medulla, in Textbook of Medical Physiology, 12th ed., Saunders Elsevier, Ed. Philadelphia, 2011, pp. 738-739
- [Background] Akselrod S, Gordon D, Ubel FA, Shannon DC, Berger AC, Cohen RJ. Power spectrum analysis of heart rate fluctuation: a quantitative probe of beat-to-beat cardiovascular control. Science. 1981 Jul 10;213(4504):220-2. doi: 10.1126/science.6166045.
- [Background] Ferrario M, Moissl U, Garzotto F, Cruz DN, Tetta C, Signorini MG, Ronco C, Grassmann A, Cerutti S, Guzzetti S. The forgotten role of central volume in low frequency oscillations of heart rate variability. PLoS One. 2015 Mar 20;10(3):e0120167. doi: 10.1371/journal.pone.0120167. eCollection 2015. PMID 25793464
- [Background] Galletly DC, Larsen PD. Relationship between cardioventilatory coupling and respiratory sinus arrhythmia. Br J Anaesth. 1998 Feb;80(2):164-8. doi: 10.1093/bja/80.2.164. PMID 9602579
- [Background] Monnet X, Rienzo M, Osman D, Anguel N, Richard C, Pinsky MR, Teboul JL. Passive leg raising predicts fluid responsiveness in the critically ill. Crit Care Med. 2006 May;34(5):1402-7. doi: 10.1097/01.CCM.0000215453.11735.06. PMID 16540963
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068